CLINICAL TRIAL: NCT05803447
Title: Analysis of Parameters Indicating the Intensity of Suicidal Behavior in Patients Suffering From Depression and Schizophrenia
Brief Title: Analysis of Parameters Indicating the Intensity of Suicidal Behavior in Psychiatric Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Other Study IDs: N/ST/ZB/17/003/3316
Record Dates: First submitted 2023-01-24; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Suicidal Behaviour; Cognitive Functions Confusion
Keywords: depression; schizophrenia; biochemical blood tests; oxidative stress pathway
MeSH Terms: conditions — Confusion; Depression; Schizophrenia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- G1K-women: The G1K group consisted of women experiencing suicidal thoughts without a tendency of implementation, in whom the result of M.I.N.I. 7.0.2 test was 1 to 8 points (n=14)
  Interventions: Other: Interview questionnaire; Diagnostic Test: biochemical parameters; Diagnostic Test: cognitive function
- G1M-men: The G1M group consisted of men experiencing suicidal thoughts without a tendency of implementation, in whom the result of M.I.N.I. 7.0.2 test was 1 to 8 points (n=16)
  Interventions: Other: Interview questionnaire; Diagnostic Test: biochemical parameters; Diagnostic Test: cognitive function
- G2K-women: The G2K group consisted of women experiencing suicidal thoughts with a tendency of implementation, in whom the result of M.I.N.I. 7.0.2 test was 9 to 16 points (n=19)
  Interventions: Other: Interview questionnaire; Diagnostic Test: biochemical parameters; Diagnostic Test: cognitive function
- G2M-men: The G2M group consisted of men experiencing suicidal thoughts with a tendency of implementation, in whom the result of M.I.N.I. 7.0.2 test was 9 to 16 points (n=9)
  Interventions: Other: Interview questionnaire; Diagnostic Test: biochemical parameters; Diagnostic Test: cognitive function
- G3K-women: The G3K group consisted of women after a suicide attempt, in whom the result of M.I.N.I. 7.0.2 test was equal to or greater than 17 points (n=15)
  Interventions: Other: Interview questionnaire; Diagnostic Test: biochemical parameters; Diagnostic Test: cognitive function
- G3M-men: The G3M group consisted of men after a suicide attempt, in whom the result of M.I.N.I. 7.0.2 test was equal to or greater than 17 points (n=17)
  Interventions: Other: Interview questionnaire; Diagnostic Test: biochemical parameters; Diagnostic Test: cognitive function
- G0K-women: The G0K group consisted of women displaying no suicidal behaviour, in whom the result of M.I.N.I. 7.0.2 test was zero points (n=10)
  Interventions: Other: Interview questionnaire; Diagnostic Test: biochemical parameters; Diagnostic Test: cognitive function
- G0M-men: The G0M group consisted of men displaying no suicidal behaviour, in whom the result of M.I.N.I. 7.0.2 test was zero points (n=20)
  Interventions: Other: Interview questionnaire; Diagnostic Test: biochemical parameters; Diagnostic Test: cognitive function

INTERVENTIONS:
Other: Interview questionnaire — An Interview questionnaire concerning an assessment of the intensity suicidal behavior, M.I.N.I. 7.0.2 was used.
  M.I.N.I. interview was conducted with each patient to verify the intensification of suicidal behaviour.
Diagnostic Test: biochemical parameters — The concentrations of the following parameters were determined from the:
  * blood serum: vitamin D3, B12, folic acid, sodium, potassium, calcium, magnesium, chlorine, total cholesterol, LDL and HDL fractions, TG
  * plasma: metabolites of the oxidative stress
Diagnostic Test: cognitive function — The participants completing cognitive function were assessed using computer CogState Test. The following cognitive functions were assessed: psychomotor drive (DET), metastability of attention (IDN), verbal memory, retrieval of learned material (ISLR) and verbal learning and memory (ISL), visual learning and memory (OCL), processing speed (GMCT), visual memory including deferred retrieval (GMR), executive functions (SETS and GML), working memory (ONB, TWOB).

SUMMARY:
The aim of this study was to analyse the level of cognitive functioning of patients with history of suicidal behaviour suffering from depression and schizophrenia, and to evaluate their oxidative stress parameters and selected biochemical parameters on the basis of bloodwork.

DETAILED DESCRIPTION:
The study was conducted among 120 patients hospitalized in the Department of Psychiatry of the UMB (Medical University of Białystok). Every participant gave their own voluntary and informed written consent. Blood parameters tests were performed in the Diagnostic Laboratory of the University's Clinical Hospital and in the Department of Hygiene, Epidemiology and Ergonomics of the Medical University of Białystok. In the first stage of the study, an M.I.N.I. 7.0.2 interview was conducted with each patient to verify the intensification of suicidal behaviour. Based on the scores, the patients were classified into one of eight groups: no suicidal behaviour group (G0K, G0M); group experiencing suicidal thoughts without a tendency of implementation (G1K, G1M); group experiencing suicidal thoughts with a tendency of implementation (G2K, G2M); group after a suicide attempt (G3K, G3M).The second stage of the study consisted of biochemical blood tests, where concentrations of vitamin D3, B12, folic acid, sodium, potassium, calcium, magnesium, chlorine, total cholesterol, LDL and HDL fractions, TG and metabolites of the oxidative stress pathway were determined. The following concentrations were determined: dityrosine (AUF/mg protein), TOS (nmol H2O2 Equiv/mg protein), TAC (umol/mg protein), OSI (TOS/TAC ratio), FRAP (μmol/mg protein), GPx (mU/mg protein), SOD (mU/mg protein) CAT (nmol H2O2/min/mg protein), AOPP (nmol/mg protein), NO (nmol/mg protein), GSH (μg/mg protein). The third stage of the study consisted of the participants completing a CogState computerized test to verify their cognitive functioning. The following cognitive functions were assessed: psychomotor drive (DET), metastability of attention (IDN), verbal memory, retrieval of learned material (ISLR) and verbal learning and memory (ISL), visual learning and memory (OCL), processing speed (GMCT), visual memory including deferred retrieval (GMR), executive functions (SETS and GML), working memory (ONB, TWOB).

ELIGIBILITY:
Inclusion Criteria:

* patients of clinical psychiatry
* patients diagnosed with schizophrenia and depression
* age: 20-50 years
* gender: women and men

Exclusion Criteria:

* exclusion criteria were any present major medical illness (somatic or neurological disease)
* use of psychoactive substances
* decreased level of cognitive functioning
* people who do not use a computer

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The research included 120 people (58 women and 62 men) who met the criteria for being incluted in the study and who did not possess exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
At the first stage, the participants were interviewed by the certified clinical psychologist. M.I.N.I. 7.0.2 interview was conducted with each patient to verify the intensification of suicidal behaviour. | in the first 48 hours after the hospital admission
  The setting of the study assumed that the procedure started in the first 48 h after the hospital admission. Based on the scores M.I.N.I.7.0.2 the patients were classified into one of eight groups:
  * control groups displaying no suicidal behaviour (G0K - women and G0M - men), the result of M.I.N.I. 7.0.2 test was zero points;
  * groups experiencing suicidal thoughts without a tendency of implementation (G1K - women and G1M - men), the result of M.I.N.I. 7.0.2 test was 1 to 8 points;
  * groups experiencing suicidal thoughts with a tendency of implementation (G2K - women and G2M - men), the result of M.I.N.I. 7.0.2 test was 9 to 16 points;
  * groups after a suicide attempt (G3K - women and G3M - men), the result of M.I.N.I. 7.0.2 test was equal to or greater than 17 points.

SECONDARY OUTCOMES:
The second stage of the study consisted of biochemical blood tests - vitamins | 1 week
  Venous blood (10 mL) was collected from all patients, then were left at room temperature for 30-60 minutes to separate the serum. After that the blood was centrifuged at 4500 x g for 20 min at 4 °C. In the next phase, some of the test tubes used to determine the concentration of vitamins (vitamin D3, B12, folic acid) were immediately used to perform these determinations standard method used in the hospital laboratory USK in Bialystok. The laboratory used Abbott equipment to perform these determinations (Architect 25-OH Vitamin D, Architect i System, Architect Follate).
The second stage of the study consisted of biochemical blood tests - ions | 1 week
  Venous blood (10 mL) was collected from all patients, then were left at room temperature for 30-60 minutes to separate the serum. After that the blood was centrifuged at 4500 x g for 20 min at 4 °C. In the next phase, some of the test tubes used to determine the concentration of ions (calcium, magnesium, chlorine, sodium, potassium) were immediately used to perform these determinations standard method used in the hospital laboratory USK in Bialystok. The laboratory used Abbott Alnity c equipment to perform these determinations. The remaining tubes were placed in a freezer at -17 to -12°C, and after 24 hours the samples were stored at the temperature of -80° C in which they were stored until being assayed (total cholesterol, LDL, HDL, TG).
The second stage of the study consisted of biochemical blood tests - total cholesterol, LDL, HDL, TG | 1 week
  Venous blood (10 mL) was collected from all patients, then were left at room temperature for 30-60 minutes to separate the serum. After that the blood was centrifuged at 4500 x g for 20 min at 4 °C. The remaining tubes were placed in a freezer at -17 to -12°C, and after 24 hours the samples were stored at the temperature of -80° C in which they were stored until being assayed (total cholesterol, LDL, HDL, TG). Total cholesterol and serum HDL cholesterol remained determined by the enzymatic-colorimetric method. The LDL cholesterol level was calculated from the formula Friedewald.
The second stage of the study consisted of biochemical blood tests - oxidative stress | 1 week
  The another laboratory tests were performer to determine parameters of oxidative stress.
  The following concentrations were determined: dityrosine (AUF/mg protein), TOS (nmol H2O2 Equiv/mg protein), TAC (umol/mg protein), OSI (TOS/TAC ratio), FRAP (µmol/mg protein), GPx (mU/mg protein), SOD (mU/mg protein) CAT (nmol H2O2/min/mg protein), AOPP (nmol/mg protein), NO (nmol/mg protein), GSH (µg/mg protein).
  The obtained plasma was precooled in liquid nitrogen and stored at -80°C. Tests were made using a Sigma-Aldrich device, using 96 well microplate reader (InfiniteM200 PROMultimode Tecan; Tecan Group Ltd) absorbance/fluorescence of the plates was measured. The results were standardized to 1 mg proteins and the measurements were performed on two samples to verify the results.

OTHER OUTCOMES:
The third stage of the study consisted of the participants completing a Cogstate (full name of the test) computerized test to verify their cognitive functioning. Part 1. | between 20 to 45 minutes
  The test was performed independently, after obtaining instructions for each task given by a psychologist. The duration of the test ranged from 20 to 45 minutes.
The third stage of the study consisted of the participants completing a Cogstate (full name of the test) computerized test to verify their cognitive functioning. Part 2. | between 20 to 45 minutes
  Parameters were evaluated using unit:
  lmn - speed of execution (log10 milliseconds) acc - accurancy (the square root of the proportion of correct answers) ter - number of errors mps - number of movements per second cor - number of correct answers err - number of errors

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ribeiro JD, Huang X, Fox KR, Franklin JC. Depression and hopelessness as risk factors for suicide ideation, attempts and death: meta-analysis of longitudinal studies. Br J Psychiatry. 2018 May;212(5):279-286. doi: 10.1192/bjp.2018.27. Epub 2018 Mar 28. PMID 29587888
- [Result] Dalglish SL, Melchior M, Younes N, Surkan PJ. Work characteristics and suicidal ideation in young adults in France. Soc Psychiatry Psychiatr Epidemiol. 2015 Apr;50(4):613-20. doi: 10.1007/s00127-014-0969-y. Epub 2014 Oct 12. PMID 25308058
- [Result] Talreja BT, Shah S, Kataria L. Cognitive function in schizophrenia and its association with socio-demographics factors. Ind Psychiatry J. 2013 Jan;22(1):47-53. doi: 10.4103/0972-6748.123619. PMID 24459374
- [Result] Kishi T, Matsuda Y, Iwata N. Memantine add-on to antipsychotic treatment for residual negative and cognitive symptoms of schizophrenia: a meta-analysis. Psychopharmacology (Berl). 2017 Jul;234(14):2113-2125. doi: 10.1007/s00213-017-4616-7. Epub 2017 May 15. PMID 28508107
- [Result] Koweszko T, Gierus J, Zalewska A, Maciejczyk M, Waszkiewicz N, Szulc A. The Relationship between Suicide and Oxidative Stress in a Group of Psychiatric Inpatients. J Clin Med. 2020 Oct 28;9(11):3462. doi: 10.3390/jcm9113462. PMID 33126414
- [Result] Roca M, Del Amo AR, Riera-Serra P, Perez-Ara MA, Castro A, Roman Juan J, Garcia-Toro M, Garcia-Pazo P, Gili M. Suicidal risk and executive functions in major depressive disorder: a study protocol. BMC Psychiatry. 2019 Aug 16;19(1):253. doi: 10.1186/s12888-019-2233-1. PMID 31420027
- [Result] Liaugaudaite V, Fineberg NA, Podlipskyte A, Gecaite J, Juskiene A, Mickuviene N, Burkauskas J. Neurocognitive markers of suicidal ideation in patients with anxiety and mood disorders. Int J Psychiatry Clin Pract. 2020 Jun;24(2):116-119. doi: 10.1080/13651501.2019.1666148. Epub 2020 Mar 12. PMID 32162978
- [Result] Yin Y, Tong J, Huang J, Tian B, Chen S, Cui Y, An H, Tan S, Wang Z, Yang F, Tian L, Tong Y, Hong LE, Tan Y. Suicidal ideation, suicide attempts, and neurocognitive dysfunctions among patients with first-episode schizophrenia. Suicide Life Threat Behav. 2020 Dec;50(6):1181-1188. doi: 10.1111/sltb.12689. Epub 2020 Sep 19. PMID 32949038
- [Result] Wang J, Tang X, Lu Y, Zheng Y, Zeng F, Shi W, Zhou P. Lycopene Regulates Dietary Dityrosine-Induced Mitochondrial-Lipid Homeostasis by Increasing Mitochondrial Complex Activity. Mol Nutr Food Res. 2022 Jan;66(1):e2100724. doi: 10.1002/mnfr.202100724. Epub 2021 Nov 28. PMID 34780105
- [Result] Moraes JB, Maes M, Roomruangwong C, Bonifacio KL, Barbosa DS, Vargas HO, Anderson G, Kubera M, Carvalho AF, Nunes SOV. In major affective disorders, early life trauma predict increased nitro-oxidative stress, lipid peroxidation and protein oxidation and recurrence of major affective disorders, suicidal behaviors and a lowered quality of life. Metab Brain Dis. 2018 Aug;33(4):1081-1096. doi: 10.1007/s11011-018-0209-3. Epub 2018 Mar 14. PMID 29542039
- [Result] Liu T, Zhong S, Liao X, Chen J, He T, Lai S, Jia Y. A Meta-Analysis of Oxidative Stress Markers in Depression. PLoS One. 2015 Oct 7;10(10):e0138904. doi: 10.1371/journal.pone.0138904. eCollection 2015. PMID 26445247
- [Result] Vergallo A, Giampietri L, Baldacci F, Volpi L, Chico L, Pagni C, Giorgi FS, Ceravolo R, Tognoni G, Siciliano G, Bonuccelli U. Oxidative Stress Assessment in Alzheimer's Disease: A Clinic Setting Study. Am J Alzheimers Dis Other Demen. 2018 Feb;33(1):35-41. doi: 10.1177/1533317517728352. Epub 2017 Sep 21. PMID 28931301
- [Result] Lang E, Lang F. Mechanisms and pathophysiological significance of eryptosis, the suicidal erythrocyte death. Semin Cell Dev Biol. 2015 Mar;39:35-42. doi: 10.1016/j.semcdb.2015.01.009. Epub 2015 Jan 28. PMID 25636585